CLINICAL TRIAL: NCT06345703
Title: A Phase 1, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and PK of Single and Multiple Ascending Oral Doses and Food Effect of NS-136 in Healthy Subjects
Brief Title: First-into-human Study of NS-136 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NeuShen Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NS136HV101; CTR20244269 (Other: China NMPA)
Record Dates: First submitted 2024-03-19; First posted 2024-04-03 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Subjects
Keywords: muscarinic m4 receptor

STUDY DESIGN:
Intervention Model Description: The trial consists of three parts: the first part is a single ascending dose (SAD) study, the second part is a multiple ascending dose (MAD) study, and the third part is food effect (FE) study. The first two parts (SAD and MAD) will be randomized, double-blind, single or multiple ascending dose and placebo-controlled study designs. The third part (FE) will be a randomized, open-label, two-period, crossover study design. To evaluate the safety, tolerability, pharmacokinetic profile, and the effect of food on the PK profile of NS-136 in healthy subjects and to determine the maximum tolerated dose (MTD)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Arm1 (Experimental): NS-136 SAD Dose 1
  Interventions: Drug: NS-136 tablet
- Arm2 (Experimental): NS-136 SAD Dose 2
  Interventions: Drug: NS-136 tablet
- Arm3 (Experimental): NS-136 SAD Dose 3
  Interventions: Drug: NS-136 tablet
- Arm4 (Experimental): NS-136 SAD Dose 4
  Interventions: Drug: NS-136 tablet
- Arm5 (Experimental): Arm5 NS-136 MAD Dose 1
  Interventions: Drug: NS-136 tablet
- Arm6 (Experimental): Arm5 NS-136 MAD Dose 2
  Interventions: Drug: NS-136 tablet
- Arm7 (Experimental): FE Grp A
  Interventions: Drug: NS-136 tablet
- Arm8 (Experimental): FE Grp B
  Interventions: Drug: NS-136 tablet
- Arm9 (Placebo Comparator): NS-136 SAD Dose 1 PBO
  Interventions: Drug: Placebo
- Arm10 (Placebo Comparator): NS-136 SAD Dose 2 PBO
  Interventions: Drug: Placebo
- Arm11 (Placebo Comparator): NS-136 SAD Dose 3 PBO
  Interventions: Drug: Placebo
- Arm12 (Placebo Comparator): NS-136 SAD Dose 4 PBO
  Interventions: Drug: Placebo
- Arm13 (Placebo Comparator): NS-136 MAD Dose 1 PBO
  Interventions: Drug: Placebo
- Arm14 (Placebo Comparator): NS-136 MAD Dose 2 PBO
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — NS-136 matching placebo
  Arms: Arm10; Arm11; Arm12; Arm13; Arm14; Arm9
Drug: NS-136 tablet — Investigational product NS-136
  Arms: Arm1; Arm2; Arm3; Arm4; Arm5; Arm6; Arm7; Arm8

SUMMARY:
The goal of this clinical trial is to exlplore the profile of NS-136 in health conditions. The main questions it aims to answer are:

* Is NS-136 safe and tolerable in heathy subjects under tested dosing regimen?
* What is the pharmacokinectic profile of NS-136 in healthy subjects under tested dosing regimen?

ELIGIBILITY:
Inclusion Criteria

Study subjects must meet all of the following criteria for study entry:

1. Healthy males or females aged 18-65 years (inclusive), with a body mass index (BMI) between 18.00 and 32.00 kg/m2(inclusive);
2. Not participated in any other clinical trials within the past 30 days or 5 half-lives of other investigational drugs prior to the screening, whichever is longer;
3. For women of reproductive potential, a negative pregnancy test is required, and they must agree to use contraception (more details see Appendix 1) from the time of signing the informed consent form until at least 90 days after the last dose of investigational product. Male subjects must agree to use adequate contraception from the time of signing the informed consent form until at least 90 days after the last dose of investigational product, and donation of sperm or ova is prohibited during the entire study period;
4. In good health, determined by the investigator on the basis of medical history, physical examinations, vital signs, 12-lead electrocardiograms (12-ECGs), clinical laboratory tests (haematology, urinalysis, blood chemistry). Repeated examination is allowed once at investigator's discretion;
5. Full understanding of the purpose, nature, procedures of the study, and the potential adverse reactions. Subject voluntarily participates and signs the informed consent form before any study procedures begin.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from study entry:

1. Individuals who are allergic to the investigational product or any of its components, or who are easily allergic at investigator's discretion;
2. Individuals who are intolerant to venipuncture/venous catheterization or blood fainting or needle phobia;
3. Positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (Anti-HCV), human immunodeficiency virus antibody (Anti-HIV) during the screening period;
4. Average daily smoking of more than 5 cigarettes in the 3 months prior to screening, or inability to stop using any tobacco products (including nicotine products) during the trial;
5. Excessive alcohol consumption or weekly alcohol intake exceeding 14 units of alcohol in the 4 weeks prior to screening (1 unit equals 10 grams of pure alcohol, alcohol content of different alcoholic beverages is indicated by volume ratio, approximately 1 alcohol unit is equal to 35 mL of 50° liquor or 350 mL of 5° beer), or unwillingness to stop drinking alcohol or consuming any products containing alcohol during the trial, or positive alcohol test upon screening and admission (repeated test is allowed once at investigator's discretion);
6. Excessive intake of tea, coffee, or caffeinated beverages (more than 8 cups/day, 1 cup = 250 mL) in the 3 months prior to screening, or inability to stop consuming any beverages or foods containing caffeine, any beverages or foods rich in purines, or grapefruit and other substances that may affect drug absorption, distribution, metabolism, or excretion during the trial;
7. History of drug abuse within the past year prior to the first dose, or positive results in a multi-drug urine screening test upon screening period and admission. Repeated test is allowed once at investigator discretion;
8. History of definite neurological or psychiatric disorders (including epilepsy, migraines, dementia, depression or bipolar disorder, schizophrenia, etc.); history of prolonged QTc interval; immunodeficiency or immunosuppressive diseases, malignant neoplastic diseases; chronic cardiovascular, hepatic, renal, endocrine, respiratory, hematological (including coagulation), digestive system diseases, cholecystectomy, Gilbert's Syndrome or resolved childhood asthma;
9. Underwent major surgery within the past 6 months prior to the first dose (such as coronary artery bypass grafting, hepatectomy, gynecological surgery, etc.); occurrence of acute neurological, digestive, respiratory, circulatory, endocrine, hematological, or other systemic diseases that may affect the absorption, distribution, metabolism, excretion, and safety evaluation of the investigational product within 3 months prior to screening judged by investigator;
10. Donated blood or experienced blood loss ≥400 mL within the 3 months prior to the first dose; difficulties in venous blood collection; planned blood donation during the study or within 1 month after the study;
11. Use of strong inhibitors or inducers of cytochrome P450 (CYP) 3A4 within 14 days prior to the administration of the investigational drug or anticipated use of strong CYP3A4 inhibitors or inducers during the study participation period;
12. Use of any prescription or non-prescription medications, including herbal and OTC medications within 14 days of dosing, with the exception of paracetamol (≤2 g per day);
13. Receipt of vaccines within the 4 weeks prior to the first dose of the investigational product;
14. Cannot tolerate high-fat meals or have special dietary requirements, or cannot adhere to a standardized diet (only for subjects in the FE trial);
15. Other factors deemed unsuitable for participation in the trial by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | for SAD, day 1-7; for MAD, day 1-26, for FE, day1-14
Main pharmacokinetic parameters | for SAD, day 1-7; for MAD, day 1-26,
  Vd/F
Main pharmacokinetic parameters | for SAD, day 1-7; for MAD, day 1-26,
  CL/F
Main pharmacokinetic parameters | for SAD, day 1-7; for MAD, day 1-26,
  t1/2
Main pharmacokinetic parameters | for SAD, day 1-7; for MAD, day 1-26,
  Tmax
Main pharmacokinetic parameters | for SAD, day 1-7; for MAD, day 1-26,
  AUC0-∞
Main pharmacokinetic parameters | for SAD, day 1-7; for MAD, day 1-26,
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Emir Redzepagic, MD, Principal Investigator — CMAX Clinical Research Pty Ltd; Xiaolan Yong Chief Pharmacist, BS, Principal Investigator — Chengdu Xinhua Hospital, China
Locations (2):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia
- Chengdu Xinhua Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet